CLINICAL TRIAL: NCT02020694
Title: The Role of Vitamin D Supplementation in the Prevention of Cardiovascular Risk Factors
Brief Title: Vitamin D Supplementation for the Prevention of Cardiovascular Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Giaccari Andrea, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 752/11; 2011-003183-75 (EudraCT Number)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Overweight; Insulin Resistance
Keywords: Obesity; Insulin resistance; Vitamin D; Cardiovascular risk factors
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vitamin D and Diet (Experimental): Cholecalciferol (vitamin D3) 25,000 I.U./2.5 mL oral solution. 25,000 I.U. (one bottle) per week.
  Hypocaloric diet
  Interventions: Drug: Vitamin D
- Placebo & Diet (Placebo Comparator): Oral solution mimicking cholecalciferol (vitamin D3) 25,000 I.U./2.5 mL. One bottle per week.
  Hypocaloric diet
  Interventions: Drug: Placebo (for vitamin D)

INTERVENTIONS:
Drug: Vitamin D
  Arms: Vitamin D and Diet
Drug: Placebo (for vitamin D)
  Arms: Placebo & Diet

SUMMARY:
Hypovitaminosis D is highly prevalent in the general population, particularly in obese individuals. Besides being associated with obesity, vitamin D deficiency seems to be involved in the pathogenesis of insulin resistance and low-grade chronic inflammation. In addition, it has been reported that individuals with low vitamin D levels are at increased risk for cardiovascular diseases. A healthy diet and weight loss are cornerstones in the prevention of cardiovascular diseases. Vitamin D supplementation could increase the beneficial effects of these lifestyle interventions. The purpose of this study is to assess whether vitamin D supplementation in conjunction with a hypocaloric diet improves the cardiometabolic profile of overweight/obese subjects to a greater extent than diet alone.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥25 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* Chronic kidney disease
* Liver disease
* Cholestasis
* Cancer
* Chronic bowel disease
* Primary or secondary hyperparathyroidism
* Treatment with drugs that may affect insulin sensitivity, weight or calcium/vitamin D metabolism
* Laxative abuse
* Changes >10% of usual body weight in the previous 6 months
* Alcohol or illicit drug abuse
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity (M value) | Baseline, 3 months
  Insulin sensitivity will be measured with the hyperinsulinemic euglycemic clamp technique and expressed as M value, calculated from the glucose infusion rate during the last 30 min of the clamp.

SECONDARY OUTCOMES:
Change from baseline in oral glucose tolerance | Baseline, 3 months
  Oral glucose tolerance will be assessed with a standard 2-hour oral glucose tolerance test (OGTT).
Change from baseline in body composition | Baseline, 3 months
  Body composition will be determined by using dual energy X-ray absorptiometry (DXA).
Change from baseline in anthropometric parameters | Baseline, 3 months
  Weight, BMI, waist and hip circumference, waist/hip ratio.
Change form baseline in systolic and diastolic blood pressure | Baseline, 3 months
Change from baseline in phosphocalcic metabolism | Baseline, 3 months
  Serum vitamin D, PTH and calcium
Change from baseline in inflammatory markers | Baseline, 3 months
  Interleukin-6 (IL-6), IL-10, adiponectin, TNF-α, C-reactive protein (CRP) and fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Giaccari, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Muscogiuri G, Policola C, Prioletta A, Sorice G, Mezza T, Lassandro A, Della Casa S, Pontecorvi A, Giaccari A. Low levels of 25(OH)D and insulin-resistance: 2 unrelated features or a cause-effect in PCOS? Clin Nutr. 2012 Aug;31(4):476-80. doi: 10.1016/j.clnu.2011.12.010. Epub 2012 Jan 20. PMID 22260937
- [Background] Muscogiuri G, Sorice GP, Prioletta A, Policola C, Della Casa S, Pontecorvi A, Giaccari A. Will vitamin D reduce insulin resistance? Still a long way to go. Am J Clin Nutr. 2011 Mar;93(3):672-3; author reply 673-4. doi: 10.3945/ajcn.110.009068. Epub 2011 Jan 5. No abstract available. PMID 21209228
- [Background] Muscogiuri G, Sorice GP, Prioletta A, Policola C, Della Casa S, Pontecorvi A, Giaccari A. Association of vitamin D with insulin resistance and beta-cell dysfunction in subjects at risk for type 2 diabetes: comment to Kayaniyil et al. Diabetes Care. 2010 Jul;33(7):e99; author reply e100. doi: 10.2337/dc10-0587. No abstract available. PMID 20587719
- [Background] Muscogiuri G, Sorice GP, Prioletta A, Policola C, Della Casa S, Pontecorvi A, Giaccari A. 25-Hydroxyvitamin D concentration correlates with insulin-sensitivity and BMI in obesity. Obesity (Silver Spring). 2010 Oct;18(10):1906-10. doi: 10.1038/oby.2010.11. Epub 2010 Feb 11. PMID 20150902
- [Derived] Cefalo CMA, Conte C, Sorice GP, Moffa S, Sun VA, Cinti F, Salomone E, Muscogiuri G, Brocchi AAG, Pontecorvi A, Mezza T, Giaccari A. Effect of Vitamin D Supplementation on Obesity-Induced Insulin Resistance: A Double-Blind, Randomized, Placebo-Controlled Trial. Obesity (Silver Spring). 2018 Apr;26(4):651-657. doi: 10.1002/oby.22132. Epub 2018 Mar 4. PMID 29504254